CLINICAL TRIAL: NCT06277453
Title: Effect of Adjuvant Chemotherapy Cycles on Patients With Node-negative Gastric Cancer Following Neoadjuvant Chemotherapy: Multicenter Cohort Study
Brief Title: Effect of Adjuvant Chemotherapy Cycles on Patients With Node-negative Gastric Cancer Following Neoadjuvant Chemotherapy
Status: Active, not recruiting | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Fujian Medical University Union Hospital, Fujian Medical University
Other Study IDs: 2024KY010
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Locally Advanced Gastric Cancer
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AC ≥5: Patients with lymph node-negative gastric cancer who received neoadjuvant chemotherapy and underwent at least five cycles of adjuvant chemotherapy (AC ≥5) after surgery
  Interventions: Other: surgery
- AC <5: Patients with lymph node-negative gastric cancer who received neoadjuvant chemotherapy and underwent at less five cycles of adjuvant chemotherapy (AC <5) after surgery
  Interventions: Other: surgery

INTERVENTIONS:
Other: surgery — radical gastric cancer surgery (R0) and D2 lymph node dissection

SUMMARY:
To explore the effect of adjuvant chemotherapy cycles on the prognosis of this specific patient with lymph node-negative gastric cancer following neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
We analyzed clinicopathological data from patients with lymph node-negative gastric cancer who underwent neoadjuvant chemotherapy at four institutions between 2010 and 2020. The 3-year OS was assessed using landmark analysis. Independent risk factors associated with 3-year OS were identified using a Cox proportional hazards regression model.

ELIGIBILITY:
Inclusion Criteria:

* (1) preoperative neoadjuvant chemotherapy; (2) primary gastric adenocarcinoma, diagnosed by gastroscopic pathology findings before neoadjuvant chemotherapy in complete pathological remission (pCR) cases or via postoperative pathology findings in all other instances; (3) absence of distant metastases in the liver, lungs, or abdominal cavity, as confirmed by preoperative chest radiography or chest computed tomography (CT), abdominal ultrasonography, abdominal CT, and other imaging; (4) radical gastric cancer surgery (R0) and D2 lymph node dissection; and (5) postoperative pathologic verification of no lymph node metastasis (i.e., lymph node-negative).

Exclusion Criteria:

* (1) preoperative radiotherapy or radiochemotherapy, (2) discovery of distant metastases preoperatively or intraoperatively, (3) coexistence of other malignant tumors, (4) residual gastric cancer, and (5) perioperative patient mortality.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with node-negative gastric cancer following neoadjuvant chemotherapy
Sampling Method: Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival | 3 years
  3-year overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Ming Huang, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Department of Gastric Surgery， Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No